CLINICAL TRIAL: NCT05076032
Title: Phase II, Randomised, Double-blind, Parallel-group, Placebo-controlled Trial to Assess Ongoing Pregnancy Rate With OXO-001 (200/300 mg) or Placebo at 10 Weeks Following Fresh Single Blastocyst Transfer From Donor Oocyte IVF/ICSI
Brief Title: Phase II Clinical Trial to Evaluate the Ongoing Pregnancy Rate With OXO-001 in IVF/ICSI With Donor Oocytes.
Acronym: OXOART2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OXOLIFE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXO-001-201; 2021-000001-25 (EudraCT Number)
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Infertility, Female; Infertility
Keywords: Endometrial receptivity; Embryo implantation
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Intervention Model Description: A phase II, randomised, double-blind, parallel-group, placebo-controlled trial to assess the ongoing pregnancy rate with OXO-001 (200 mg, 300 mg) or placebo at 10 weeks following fresh single blastocyst transfer resulting from donor oocyte IVF/ICSI.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OXO-001 200 mg (Experimental): Two tablets of 100 mg have to be taken once daily in the early morning.
  Interventions: Drug: OXO-001
- OXO-001 300 mg (Experimental): Two tablets of 150 mg have to be taken once daily in the early morning.
  Interventions: Drug: OXO-001
- Placebo (Placebo Comparator): Two tablets have to be taken once daily in the early morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OXO-001 — OXO-001 oral administration once daily in the early morning. The treatment duration will vary depending on the woman, but it will last between 10 to 14 weeks approximately.
  Arms: OXO-001 200 mg; OXO-001 300 mg
Drug: Placebo — Placebo oral administration once daily in the early morning. The treatment duration will vary depending on the woman, but it will last between 10 to 14 weeks, approximately.
  Arms: Placebo

SUMMARY:
The main objective of this clinical research trial is to test the efficacy of OXO-001 in a daily oral administration increasing the pregnancy rate in IVF/ICSI by preparing the uterus to receive the embryo.

DETAILED DESCRIPTION:
Assisted reproductive techniques are the most common procedures to fulfill the desire for pregnancy in infertile women. Unfortunately, more than half of the assisted reproduction cycles result in implantation failure or early pregnancy loss, the two main causes of infertility and the most important unmet medical need in the field of infertility with current treatments.

This clinical trial aims to test the capacity of OXO-001 to enhance embryo implantation. It is a phase II, randomised, double-blind, parallel-group, placebo-controlled trial that will assess the ongoing pregnancy rate with OXO-001 (200 mg, 300 mg) or placebo at 10 weeks following fresh single blastocyst transfer resulting from donor oocyte IVF/ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent.
* Infertile female subjects indicated for egg donor programme in the context of ART.
* Subjects aged ≥ 18 to ≤ 45 years at screening.
* Body mass index (BMI) ≥ 18.0 and < 30.0 kg/m2.
* Normal results of a 2-dimensional (2D) or 3-dimensional (3D) transvaginal US (TVUS) at screening.
* Planned transfer of a fresh single blastocyst from a donated egg.
* Good quality sperm.
* Planned endometrial preparation and luteal support.

Exclusion Criteria:

* History of two or more failed in-vitro fertilisation (IVF) / intra-cytoplasmic sperm injection (ICSI) cycles after embryo transfer of donor oocyte during the last attempts prior to the trial.
* Gynaecological abnormality relevant to the ART procedure and outcome, which in the opinion of the investigator could interfere with the trial objectives.
* Abnormal haemorrhage of the reproductive tract of undetermined origin.
* Endometrial biopsy or endometrial local injury within one month prior to screening.
* Diagnosis of severe endometriosis and/or adenomyosis.
* Positive hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus results.
* Relevant clinically significant abnormality in the results of safety laboratory tests at screening.
* Systemic disease which might interfere with the purpose of the trial.
* Any malignant neoplasm.
* Known history of venous thrombosis or thromboembolism, including any coagulation abnormality leading to an increased risk of clotting.
* History of uncontrolled hypertension.
* Known hypersensitivity to any component of the IP used in this trial.
* Known allergy, hypersensitivity or any other contraindications to preparations used in the context of endometrial preparation and fresh ET with a donated egg.
* History (within 12 months) of or known current problems with alcohol or substance abuse.
* Any condition or treatment that, in the opinion of the investigator, may jeopardise the trial conduct according to the protocol.
* Previous treatment with the IP of this trial at any time or participation in another clinical trial within the past 3 months prior to screening.
* Employees of the investigator or trial centre, with direct involvement in the proposed trial or other studies under the direction of that investigator or trial centre, as well as family members of the employees or the principal investigator.
* Persons committed to an institution by virtue of an order issued either by the judicial or other authorities.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 408 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10 weeks post Embryo Transfer (ET)
  Rate of subjects with uterine pregnancy and a foetal heartbeat confirmed by ultrasound (US)

SECONDARY OUTCOMES:
Positive blood pregnancy test | 10 to 15 days post ET
  Percentage of women with positive blood pregnancy test
Vital pregnancy at 6 weeks | 6 weeks post ET
  Intra-uterine pregnancy with foetal heartbeat at 6 weeks post ET
Early pregnancy loss rate | 10 weeks post ET
  Early pregnancy loss rate within 10 weeks of gestation (i.e. after positive blood pregnancy test 10-15 days post ET).
Adverse events | From the first intake of the investigational product until 10 weeks post ET
  Incidence and severity of adverse events/serious adverse events
Hematology and biochemistry values | From the first intake of the investigational product until 10 weeks post ET
  Changes from baseline in haematology and biochemistry values
Vital signs | From the first intake of the investigational product until 10 weeks post ET
  Changes from baseline in heart rate (bpm)
Vital signs | From the first intake of the investigational product until 10 weeks post ET
  Changes from baseline blood pressure mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Arbat, MD, Study Director — Oxolife S.L
Locations (28):
- Czechia (7):
  - Fertimed s.r.o., Olomouc
  - ISCARE centrum asistované reprodukce, Prague
  - IVF CUBE, Prague
  - Sanatorium PRONATAL, Prague
  - UNICA Prague s.r.o, Prague
  - Pronatal NORD, Teplice
  - Klinika reprodukční medicíny a gynekologie, Zlín
- Poland (6):
  - KRIOBANK Centrum Leczenia Niepłodności Ginekologia, Bialystok
  - ProCrea Swiss IVF Center s.r.o., Katowice
  - Provita Sp. z o.o., Katowice
  - VitroLive Sp. z o.o., Szczecin
  - OVIklinika, Warsaw
  - Przychodnia Lekarska nOvum, Katarzyna Kozioł, Piotr Lewandowski spółka jawna, Warsaw
- Spain (15):
  - Instituto Bernabeu, Alicante
  - Fertty, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitario Quirónsalud Barcelona, Barcelona
  - IVI Barcelona, Barcelona
  - IVI Bilbao, Leioa
  - GINEFIV Madrid, Madrid
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Instituto Bernabeu Madrid, Madrid
  - IVI Madrid, Madrid
  - IVI Mallorca, Palma de Mallorca
  - Ginemed Sevilla, Seville
  - IVI Sevilla, Seville
  - IVI Valencia, Valencia
  - IVI Zaragoza, Zaragoza